CLINICAL TRIAL: NCT01814527
Title: High Dose Omega-3 Fatty Acids in the Treatment of Sport Related Concussions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, David Bica DO, Clinical Assistant Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DSM-2012-1059
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Results first posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Mild Concussion; Brain Concussion; Cerebral Concussion
Keywords: Fish oil; Omega 3 Fatty acids; Docosahexaenoic acid; Mild Concussion; Brain Concussion; Cerebral Concussion
MeSH Terms: conditions — Brain Concussion | interventions — Docosahexaenoic Acids; Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docosahexaenoic acid (Active Comparator): The experimental group will be given a standardized dose of omega-3 fatty acid containing 2200mg of DHA for 30 days after onset of concussion or longer for those with continued symptomatology. Brain Armor an over the counter DHA supplements that is independently tested and certified by the National Science Foundation Athletic Banned Substance Certified for Sport Program. The Docosahexaenoic acid supplement has 440mg of DHA per capsule and each subject will be given 5 capsules of Brain Armor once daily for a DHA dose of 2200mg/day.
  Interventions: Dietary Supplement: Docosahexaenoic acid
- Placebo (Placebo Comparator): The placebo group will be given an equal amount of capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Docosahexaenoic acid — 5 capsules containing 440mg of Docosahexaenoic acid (DHA)for total daily dosing of 2200mg of DHA daily
  Other Names: Omega-3 Fatty Acids
  Arms: Docosahexaenoic acid
Drug: Placebo — 5 capsules that are identical to the treatment.
  Arms: Placebo

SUMMARY:
Concussions are defined as a complex pathophysiological process affecting the brain, induced by traumatic biomechanical forces. Currently the standard of care in the treatment for concussions is cognitive and physical rest until symptoms resolve with a graduated return to activity. High dose omega-3 fatty acids have shown to have anti-inflammatory, anti-oxidant, and membrane stabilizing properties. They have also been used in treatment of severe traumatic brain injury. The purpose of this study is to determine if early high dose omega-3 fatty acid supplementation in Division I National Collegiate Athletic Association (NCAA) athletes that have sustained a concussion will decrease the number of days out of competitive sports with a quicker symptom resolution, return to baseline neurocognitive functioning and postural stability using a randomized double blind placebo controlled study design. Once an athlete is identified as having sustained a concussion by the East Carolina University Sports Medicine staff and qualifies for the study, he/she will randomly be assigned to either high dose omega-3 fatty acid or placebo. Both groups will undergo standard and usual care for concussed athletes at East Carolina University. The number of days it takes the athlete to return to competitive athletics will be recorded, along with time to symptom resolution, normalization of their computerized neurocognitive testing (ImPact) and computerized postural stability testing (Biodex BioSway).

DETAILED DESCRIPTION:
In the United States, an estimated 1.7 million people sustain a traumatic brain injury (TBI) annually; associated with 1.365 million emergency room visits and 275,000 hospitalizations annually with associated direct and indirect cost estimated to have been 4 billion in the United States in 2000. Furthermore, the US Center for Disease Control and Prevention estimates that 1.6 to 3.8 million concussions occur in sports and recreational activities annually.3 However, these figures grossly underestimate the total burden of traumatic brain injuries (TBIs) and concussions, because many individuals suffering from mild to moderate TBIs do not seek medical attention.

Even though concussion is a type of TBI that has been frequently used interchangeably with mild TBI in the medical literature; mild refers to the initial impact rather than the long-term sequelae from the injury. Historically, the definition of concussion has not been well defined, until the 3rd International Conference on Concussion in Sport (Zurich 2008) defined concussion as a complex pathophysiological process affecting the brain, induced by traumatic biomechanical forces. Several common features that incorporate clinical, pathological and biomechanical injury constructs that may be utilized in defining the nature of concussive head injury include: Concussion may be caused either by a direct blow to the head, face, neck or elsewhere on the body with an "impulsive" force transmitted to the head. This injury typically results in the rapid onset of short-lived impairment of neurologic function that resolves spontaneously. It may result in neuropathological changes, but the acute clinical symptoms largely reflect a functional disturbance rather than a structural injury. It results in a graded set of clinical signs and symptoms that may or may not involve loss of consciousness. Resolution of the clinical and cognitive symptoms typically follows a sequential course; however, it is important to note that, in a small percentage of cases, post-concussive symptoms may be prolonged. No abnormality on standard structural neuro-imaging studies is seen in concussion. Current data shows that on average 91% of athletes who sustain a concussion have their symptoms and cognitive impairment resolved in 7 ± 1.5 days and balance deficits resolved by day 5.13 Currently the main treatment for concussion is cognitive and physical rest until symptoms resolve with a graduated return to activity.

The neuropathological changes after a concussion result in functional disturbances and the clinical syndrome results from the depolarization and potassium efflux from neurons that trigger the release of excitatory amino-acids like glutamine, which in turn activate N-methyl-D-aspartate (NMDA) receptors and form a pore through which calcium enters the neuron. A large influx of calcium into the cell triggers the lysis of arachidonic acid, calpain activation and initiation of apoptosis, and the formation of reactive oxygen species (ROS). Studies have shown that the incorporation of omega-3 fatty acids into the cell membrane has been associated with decreased generation of intracellular ROS and consequent diminished activation of redox-sensitive transcription factors, such as the nuclear factor- κβ system, modifying the expression of pro-inflammatory genes. Incorporation of omega-3 fatty acids also appears to alter the properties of lipid rafts and caveolae, contributing to membrane fluidity, hormone-receptor binding and the function of membrane associated proteins are affected. Omega-3 fatty acids are also associated with decreased levels of markers and mediators of inflammation such as the cytokines interleukin-1β and tumor necrosis factor (TNF-α).

Mills et al looked at the effects of omega-3 fatty acid supplementation in a head injury model in rats. Docosahexaenoic acid (DHA) was started approximately 24 hours after injury, in the following doses: 10 mg/kg/day for group 1 and 40 mg/kg/day for group 2. The number of beta-amyloid precursor protein (APP)-positive axons was used to measure the level of injury. There was a significant quantitative difference of 182 ± 44.6 APP-positive axons in un-supplemented animals versus sham-injured animals (control animals), which had 4.1 ± 1.3 APP-positive axons per square millimeter. Group 1 showed 26.1 ± 5.3 and group 2 showed 19.6 ± 4.7, APP-positive axons. It is notable that the omega-3 fatty acid supplementation groups had a significantly reduced number of APP-positive axons at 30 days after injury to levels similar to those in uninjured animals. This study shows pathologic improvement with high dose omega-3 fatty acid supplementation, specifically DHA, in a head injury rat model. However, there are no current human studies in the medical literature that look at omega-3 fatty acid supplementation in the treatment of concussions. Does high dose omega-3 fatty acid supplementation in Division I NCAA athletes that have sustained a concussion improve time to symptom resolution, neurocognition and postural stability and thus decrease the number of days out of competitive sports? Protocol: Once an athlete qualifies for the study he/she will be randomly be assigned to either high dose omega-3 fatty acid/DHA supplementation or placebo. Demographics of the athlete will be obtained which include: age, gender, sport, academic year, height, weight, BMI, history of prior concussion, migraines, learning disability, or psychiatric diagnosis. Both groups will undergo standard and usual care for concussed athletes at East Carolina University. The physician and the athletic training staff evaluating and clearing the athlete to return to activity will be blinded.

Currently East Carolina University employs a regimented return-to-play protocol for every student-athlete that has sustained a concussion. As part of their pre-participation physical, all student-athletes will have a baseline computerized postural stability test using Biodex BioSway and a computerized neurocognitive test using ImPact. At the time of injury a Sport Concussion Assessment Tool 2 (SCAT2) is administered by a certified athletic trainer, and the student-athlete is withdrawn from participation if they are symptomatic and/or have deficits noted. The same day a concussion is suspected a repeat Biodex postural stability test will also be administered and the student-athlete is given a detailed information sheet on instructions for monitoring and follow-up. A repeat Impact neurocognitive test will then be administered within 24 hours after the injury. The student-athlete is then seen and examined by a sports medicine physician to review the results, perform a clinical exam and confirm the diagnosis. The student-athlete is then evaluated daily with a modified Symptom Evaluation Questionnaire found on the SCAT2 by an athletic trainer. When the student-athlete is asymptomatic with activities of daily living (ADLs) for 24 hours, he/she then begins a non-contact return to play protocol resembling Zurich's beginning with a supervised cardiovascular challenge. This includes 30 minutes of supervised light aerobic activity on a treadmill or stationary bike. If the athlete is asymptomatic with the cardiovascular challenge then he/she can progress to noncontact sport specific drills the subsequent day. If the athlete is still doing well he/she can progress their non-contact training drills and start light resistance training the following day. If the student-athlete remains asymptomatic through the non-contact activity progression, he/she then re-takes the computerized neurocognitive test, postural stability assessment and is re-evaluated by the physician. If the postural stability assessment and neurocognitive test are back to baseline the athlete is then cleared at the discretion of the treating sports medicine physician to return to full unrestricted activity. However, if a student-athlete's symptoms continue by day 7 both Impact and Biodex BioSway evaluation will be re-administered. This will be repeated again at 14 days and 30 days post-injury if the student-athlete continues to be symptomatic.

ELIGIBILITY:
Inclusion Criteria:

1. East Carolina University NCAA Division I athlete.
2. Have sustained a concussion within the past 24 hours.
3. A neurological exam not consistent with concern for an intracranial hemorrhage or other significant pathology.
4. Must be at least 18 years old.

Exclusion Criteria:

1. Subjects with a recent prior concussion within the past 30 days.
2. Subjects with a history of moderate to severe TBI that has required hospitalization or resulted in prolonged signs and/or symptoms (>3 weeks).
3. Subjects with a known neurological diagnosis associated with impaired cognitive function other than Attention Deficit Hyperactive Disorder or Attention Deficit Disorder.
4. Subjects already routinely using omega-3/DHA supplementation.
5. Subjects with a known allergy to algae, omega-3 fatty acid, or any component of the formulation.
6. Subjects currently requiring anticoagulants (ie: Warfarin), anti-platelets (ie: aspirin, Plavix) or any Non-steroidal anti-inflammatory drugs (ie: Ibuprofen, Naprosyn).
7. Subjects with known liver pathology or significantly elevated liver function tests (greater than 3 x normal).
8. Subjects with a current lower extremity injury that will affect postural stability testing.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P Bica, DO, Principal Investigator — East Carolina University; Joseph Armen, DO, Principal Investigator — East Carolina University
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data in collection phase and not ready for analysis

REFERENCES:
- [Background] Langlois JA, Rutland-Brown W, Wald MM. The epidemiology and impact of traumatic brain injury: a brief overview. J Head Trauma Rehabil. 2006 Sep-Oct;21(5):375-8. doi: 10.1097/00001199-200609000-00001. PMID 16983222
- [Background] McCrory P, Meeuwisse W, Johnston K, Dvorak J, Aubry M, Molloy M, Cantu R. Consensus statement on concussion in sport - The 3rd international conference on concussion in sport held in Zurich, November 2008. PM R. 2009 May;1(5):406-20. doi: 10.1016/j.pmrj.2009.03.010. No abstract available. PMID 19627927
- [Background] Giza CC, Hovda DA. The Neurometabolic Cascade of Concussion. J Athl Train. 2001 Sep;36(3):228-235. PMID 12937489
- [Background] Ma DW, Seo J, Davidson LA, Callaway ES, Fan YY, Lupton JR, Chapkin RS. n-3 PUFA alter caveolae lipid composition and resident protein localization in mouse colon. FASEB J. 2004 Jun;18(9):1040-2. doi: 10.1096/fj.03-1430fje. Epub 2004 Apr 14. PMID 15084525
- [Background] Li Q, Wang M, Tan L, Wang C, Ma J, Li N, Li Y, Xu G, Li J. Docosahexaenoic acid changes lipid composition and interleukin-2 receptor signaling in membrane rafts. J Lipid Res. 2005 Sep;46(9):1904-13. doi: 10.1194/jlr.M500033-JLR200. Epub 2005 Jun 1. PMID 15930520
- [Background] Massaro M, Habib A, Lubrano L, Del Turco S, Lazzerini G, Bourcier T, Weksler BB, De Caterina R. The omega-3 fatty acid docosahexaenoate attenuates endothelial cyclooxygenase-2 induction through both NADP(H) oxidase and PKC epsilon inhibition. Proc Natl Acad Sci U S A. 2006 Oct 10;103(41):15184-9. doi: 10.1073/pnas.0510086103. Epub 2006 Oct 3. PMID 17018645
- [Background] Massaro M, Basta G, Lazzerini G, Carluccio MA, Bosetti F, Solaini G, Visioli F, Paolicchi A, De Caterina R. Quenching of intracellular ROS generation as a mechanism for oleate-induced reduction of endothelial activation and early atherogenesis. Thromb Haemost. 2002 Aug;88(2):335-44. PMID 12195709
- [Background] Endres S, Ghorbani R, Kelley VE, Georgilis K, Lonnemann G, van der Meer JW, Cannon JG, Rogers TS, Klempner MS, Weber PC, et al. The effect of dietary supplementation with n-3 polyunsaturated fatty acids on the synthesis of interleukin-1 and tumor necrosis factor by mononuclear cells. N Engl J Med. 1989 Feb 2;320(5):265-71. doi: 10.1056/NEJM198902023200501. PMID 2783477
- [Background] Calder PC. Immunomodulation by omega-3 fatty acids. Prostaglandins Leukot Essent Fatty Acids. 2007 Nov-Dec;77(5-6):327-35. doi: 10.1016/j.plefa.2007.10.015. Epub 2007 Nov 26. PMID 18032006
- [Background] Mills JD, Bailes JE, Sedney CL, Hutchins H, Sears B. Omega-3 fatty acid supplementation and reduction of traumatic axonal injury in a rodent head injury model. J Neurosurg. 2011 Jan;114(1):77-84. doi: 10.3171/2010.5.JNS08914. Epub 2010 Jul 16. PMID 20635852
- [Background] McCrea M, Guskiewicz KM, Marshall SW, Barr W, Randolph C, Cantu RC, Onate JA, Yang J, Kelly JP. Acute effects and recovery time following concussion in collegiate football players: the NCAA Concussion Study. JAMA. 2003 Nov 19;290(19):2556-63. doi: 10.1001/jama.290.19.2556. PMID 14625332
- [Derived] Lucke-Wold B, Zasler ND, Ruchika F, Weisman S, Le D, Brunicardi J, Kong I, Ghumman H, Persad S, Mahan D, Delawan M, Shah S, Aghili-Mehrizi S. Supplement and nutraceutical therapy in traumatic brain injury. Nutr Neurosci. 2025 Jun;28(6):709-743. doi: 10.1080/1028415X.2024.2404782. Epub 2024 Dec 30. PMID 40440029

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 62 NCAA Division I Student Athletes were recruited during the 2013-2017 academic years.
Period: Overall Study
Arm/Group | Docosahexaenoic Acid | Placebo
Started | 29 | 33
Completed | 23 | 32
Not Completed | 6 | 1
Not completed — RTP greater than 30 days | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Docosahexaenoic Acid | Placebo | Total
Number analyzed (Participants) | 23 | 32 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 32 | 55
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.7 (1.4) | 19.9 (1.4) | 19.8 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 14 | 19 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 32 | 55
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.7 (6.1) | 28.3 (6.1) | 28 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Days to Return to Full Unrestricted Athletic Participation
Description: Primary outcome will be the total number of days from onset of concussion it takes for the athlete to return to unrestricted full participation in their respective sport.
Time Frame: 30 days
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Docosahexaenoic Acid | Placebo
Number analyzed (Participants) | 23 | 32
Days | 11.0 [9.1 to 13.0] | 11.9 [10.0 to 13.8]

ADVERSE EVENTS:
Time Frame: 30 days
Description: 0
Arm/Group | Docosahexaenoic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/32
Other Adverse Events (participants affected / at risk) | 0/23 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-04-25): https://cdn.clinicaltrials.gov/large-docs/27/NCT01814527/Prot_SAP_ICF_000.pdf